CLINICAL TRIAL: NCT06489223
Title: Study of Acceptability and Tolerance of an Orofacial Myofunctional Rehabilitation Pacifier in Infants
Acronym: YooTET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL23_0811
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Obstructive Sleep Apnea Syndrome; pacifier
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Use of an Orofacial Myofunctional Rehabilitation Pacifier (Experimental): The device will be offered to the child during waking periods during three tests which will be programmed remotely or not from a bottle. Each of this tests will last 15 minutes. Tests taking place near a meal must take place within 20 minutes before or after the bottle. The last test will be offered at bedtime with the aim of the child falling asleep with the device.
  Interventions: Device: Orofacial Myofunctional Rehabilitation Pacifier

INTERVENTIONS:
Device: Orofacial Myofunctional Rehabilitation Pacifier — The pacifier will be offered to the child

SUMMARY:
The development of the medical device tested was inspired by palatal plates used to treat myofunctional disorders in young patients with Down syndrome.

This protocol is intended to evaluate the acceptability and tolerance of this pacifier in infants aged 1 to 6 months during 4 test.

If acceptability and tolerance are satisfactory, an effectiveness study will be carried out to determine whether this medical device could prove useful in preventing the occurrence of Obstructive Sleep Apnea Syndrome (OSAS) in very young children, via orofacial myofunctional rehabilitation

ELIGIBILITY:
Inclusion Criteria:

* Infant aged 4 weeks to 6 months coming to the pediatric sleep department to perform a polysomnography or polygraphy with video, during hospitalization of at least 24 hours,
* Affiliate or beneficiary of a social security scheme,
* With informed consent of the 2 legal representatives.

Exclusion Criteria:

* Known allergy to silicone.

Ages: 4 Weeks to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
assess the acceptability of the pacifier in the mouth while awake | Day 1 inclusion
  cumulative time during which the pacifier is kept in the mouth over three 15-minute sessions of awake testing. The pacifier will be judged as accepted if at least 15 minutes of pacifier in the mouth are accumulated over the 3 tests carried out.

SECONDARY OUTCOMES:
Evaluate the attitude of infants when taking the pacifier in the mouth | Day 1 inclusion
  presence of grimaces when offering the pacifier in the mouth or non-nutritive sucking behavior during each test
Evaluate whether the pacifier is held in the mouth while awake | Day 1 inclusion
  Number of times the child rejects the pacifier and the maximum duration of uninterrupted hold in the mouth during the 15 minutes of each test
Evaluate how well the pacifier stays in the mouth during sleep | Day 1 inclusion, during the night
  Time during which the pacifier is kept in the mouth during sleep until spontaneous rejection, measured from a video recording, correlated to the parameters recorded by polysomnography (sleep efficiency, apnea-hypopnea index, number of microphones -arousals, total sleep time and sleep latency).
Assessment of the safety of the pacifier in infants | Day 1 inclusion
  Recording of any adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Patricia FRANCO, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Sleep pediatric unit , Woman Mother Child Hospital, Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No